CLINICAL TRIAL: NCT06441422
Title: Effectiveness of Low Load Resistance Training With Blood Flow Restriction in Individuals With Disabilities
Brief Title: Blood Flow Restriction Training for People With Disabilities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Beth Weinman, Assistant Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO00051215
Record Dates: First submitted 2024-05-20; First posted 2024-06-04 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Weakness, Muscle
Keywords: Disability; Blood flow restriction; Low load blood flow restriction training
MeSH Terms: conditions — Muscle Weakness | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low load resistance training with blood flow restriction (Experimental): Low load resistance training routine at 30-50% of a person's 1-repetition maximum with arterial occlusion pressure at 80%
  Interventions: Other: Blood flow restriction training
- Low load resistance training (Active Comparator): Low load resistance training routine at 30-50% of a person's 1-repetition maximum
  Interventions: Other: No blood flow restriction training

INTERVENTIONS:
Other: Blood flow restriction training — Participants randomized to blood flow restriction training will complete low load resistance training exercises while the limb is occluded at 80% arterial occlusion pressure.
  Arms: Low load resistance training with blood flow restriction
Other: No blood flow restriction training — Participants randomized to no blood flow restriction training will complete low load resistance without occlusion.
  Arms: Low load resistance training

SUMMARY:
A large portion of the American population live with disabilities. People with disabilities can find it difficult to perform standard exercise routines. Regular exercise is necessary to be healthy, especially as people age. Lack of exercise can lead to secondary health concerns, like loss of muscle mass, diabetes, heart attack or stroke, to name a few. For exercise to be most beneficial, a certain degree of intensity must be achieved. Low load blood flow restriction training may be able to mimic the intensity of beneficial exercise without actually exercising hard. It may be a good option for people with disabilities who find it difficult to exercise.

DETAILED DESCRIPTION:
A significant portion of the American population currently lives with a disability. There are about 300,000 Americans living with a spinal cord injury (SCI) with approximately 18,000 new cases each year. Cerebrovascular accidents (CVA), or strokes, occur at 795,000 new cases per year in the USA with strokes being the third-leading cause of death and disability combined in the world3. There are about 750,000 US adults living with multiple sclerosis (MS), 30,000 US adults with ALS, about 1400 Americans are born each year with spina bifida, about 11,000 Americans are born each year with cerebral palsy, and there were 1.6 million American amputees as of 2005, with that number expected to double by 2050. These disabilities tend to reduce the activity levels of these individuals, which puts them at an increased risk of developing comorbidities such as obesity, insulin resistance, dyslipidemia, and more. These comorbidities are often already present in those who have had a CVA, and those who are older experience an even greater burden than those who are younger. Thus, exercise regimens are crucial to maintaining their health.

Aging is associated with an increase in susceptibility to injury and a decrease in functional ability related to a decrease in muscle size and strength. This age-related decrease is also known as primary sarcopenia. Resistance exercise, such as weightlifting, has been shown to improve muscle size and strength and functional ability in elderly individuals, and resistance exercise is widely regarded as the best method to slow the progression of primary sarcopenia. Resistance exercise and physical activity has also been shown to reduce the odds of developing sarcopenia later in life, suggesting an impetus for beginning an exercise regimen while young, though any age will benefit.

Blood flow restriction (BFR) training is a method of exercise that involves restricting the participant's blood flow to the target muscle group during exercise. Historically, training to increase muscle thickness and strength occurs at 70% of a person's 1 repetition maximum (1RM), which is the maximum weight someone can lift in one repetition (rep) of a given exercise. For example, if someone's 1RM for barbell biceps curl is 100lbs, he could train at 70lbs for 3 sets of 8-12 to increase his biceps curl 1RM and the size of his biceps. This training is hereto referred as high intensity resistance training (HLRT). Training at 30-50% 1RM with BFR, hereto referred as low load blood flow restriction training (LLBFR), increases muscle thickness similar to training at 50-80% 1RM without BFR. This also results in an increase in strength due to the increase in overall muscle mass. LLBFR training regimens also display greater increases in muscle size and strength when compared to identical exercise regimens but without BFR. So, training barbell biceps curl at 30-50lbs with blood flow restriction will increase biceps size similarly to our HLRT example. It will increase biceps strength too, but likely not to the same degree as our HLRT example. However, the increase in biceps strength and size in this LLBFR example will be greater than if this person trained at 30-50lbs but without BFR. Thus, LLBFR can induce similar benefits to traditional HLRT but with a much lighter load.

Due to the efficacy and efficiency of LLBFR in increasing muscle size and strength, it has been proposed as an alternate exercise regimen for those unable to tolerate, or are contraindicated for, traditional HLRT, such as the elderly or individuals with disabilities. This study proposes to examine if LLBFR is beneficial when compared to traditional low load resistance training.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age > or = 18
* English speaking
* Able to understand and perform upper extremity exercises

Exclusion Criteria:

* Pregnant
* Body mass index >40 kg·m-2
* Uncontrolled hypertension (>150/90 mmHg)
* Presence of neuromuscular junction and other muscle diseases
* Myocardial infarction in the past 6 months
* Unstable cardiovascular disease
* History of an upper limb deep vein thrombosis
* History of autonomic dysreflexia
* Upper extremity fracture within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in strength between low load blood flow restriction resistance training and low load resistance training | 6 weeks
  This outcome will measure the efficacy of low load blood flow restriction training (LLBFR) on muscle strength. The difference in muscle strength as measured by change in 1-repetition maximum weight in pounds will be compared in individuals training with LLBFR on their arm extensors and individuals training with low load resistance training (LLRT) on their arm extensors compared to their baseline.
Difference in arm circumference between low load blood flow restriction resistance training and low load resistance training | 6 weeks
  This outcome will measure the efficacy of low load blood flow restriction training (LLBFR) on arm circumference. The difference in arm circumference as measured by tape measure will be the change in centimeters in individuals training with LLBFR on their arm extensors compared to individuals training with low load resistance training (LLRT) on their arm extensors when compared to their respective baseline.
Difference in muscle thickness change between low load blood flow restriction resistance training and low load resistance training | 6 weeks
  This outcome will measure the efficacy of low load blood flow restriction training (LLBFR) on muscle thickness. The difference in muscle thickness as measured by ultrasound will be the change in centimeters in individuals training with LLBFR on their arm extensors compared to individuals training with low load resistance training (LLRT) on their arm extensors when compared to their respective baseline.

SECONDARY OUTCOMES:
The interaction effect between disability status (disable versus able-bodied) and training group (LLBFR and LLRT) on the change in strength. | 6 weeks
  Response to training in individuals with disabilities. The results of LLBFR on muscle strength as measured by change in pounds of 1-repetition maximum to the arm extensors will be compared between those with disabilities and those without.
The interaction effect between disability status (disable versus able-bodied) and training group (LLBFR and LLRT) on the change in arm circumference. | 6 weeks
  Response to training in individuals with disabilities. The results of LLBFR on arm circumference as measured by change in centimeters as measured by tape measure to the arm extensors will be compared between those with disabilities and those without.
The interaction effect between disability status (disable versus able-bodied) and training group (LLBFR and LLRT) on the change in muscle thickness. | 6 weeks
  Response to training in individuals with disabilities. The results of LLBFR on muscle thickness as measured by ultrasound in change in centimeters to the muscle thickness will be compared between those with disabilities and those without.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No